CLINICAL TRIAL: NCT01564225
Title: A Phase 1, Open-label, Multicenter, Safety and Pharmacokinetic Study of EDI200, an Ectodysplasin-A1 Replacement Molecule, in X-Linked Hypohidrotic Ectodermal Dysplasia (XLHED) Adults
Brief Title: A Phase 1, Open-label, Multicenter, Safety and Pharmacokinetic Study of EDI200
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Edimer Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECP-004
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: X-linked Hypohidrotic Ectodermal Dysplasia
Keywords: XLHED
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic | interventions — Fc-EDA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EDI200 (Experimental)
  Interventions: Drug: EDI200

INTERVENTIONS:
Drug: EDI200 — Cohort 1 will be dosed at 3 mg/kg/dose. Cohort 2 will be dosed at 10 mg/kg/dose. Both cohorts will receive 2 doses/week for a total of 5 doses.

SUMMARY:
Following discussions with the FDA, a Phase 1 safety study is being initiated in X-Linked Hypohidrotic Ectodermal Dysplasia (XLHED)-affected adults to develop safety and exposure data for EDI200 in anticipation of dosing XLHED-affected neonates. Selecting XLHED-affected adults for this study provides a genetic match and biologic relevance to XLHED-affected neonates. Both males and females will be enrolled, providing safety experience with EDI200 that will inform the planned neonate study as well as supportive data for potential future trials of antenatal EDI200 administration.

DETAILED DESCRIPTION:
The Phase 1 study will enroll two cohorts of 3 XLHED-affected adults each, for a total of 6 subjects. The size and scope of the study design are consistent with a drug development program in an ultra-rare disease and supported by the absence of safety concerns in a GLP non-human primate toxicology study. All subjects must meet entry criteria including documentation of an EDA mutation. Mirroring the conditions of use anticipated for the XLHED-affected newborn study, the adult cohort study incorporates a multiple-dose regimen associated with maximal efficacy in the newborn canine model. Primary outcome measures will be safety, tolerability, immunogenicity and pharmacokinetics (PK). While current data does not support a likelihood of clinical benefit for the XLHED-affected adult subjects, assays of pharmacodynamic/biologic activity are incorporated into the study design as exploratory objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of child-bearing age, age 18-40 years
2. Weight between 45 and 90 kg and a body mass index (BMI) from 18 to 29 kg/m2 (calculated using the following formula: weight in kilograms/(height in meters)2)
3. Both males and females must be documented (via genetic testing) to carry an EDA mutation associated with XLHED; or have the clinical signs and symptoms associated with HED and/or a family history of HED and provide a blood sample to be sent for genetic testing that confirms an EDA mutation associated with XLHED
4. No major medical issues that the investigator considers to be a contraindication of participation
5. No scalp shaving in the month prior to first dose (males only)
6. Women must use a "highly effective" method of contraception throughout the trial. Highly effective methods of birth control are defined as those, alone or in combination, which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly. These methods include implants, injectables, oral contraceptives, some intrauterine contraceptive devices, sexual abstinence, tubal ligation or a vasectomized partner.
7. No treatment with an investigational drug within the last three months
8. Signed written informed consent

Exclusion Criteria:

1. Women who are pregnant (confirmed via urine pregnancy test) or breastfeeding at screening or planning to become pregnant at any time during the study period
2. Known history of hepatitis B surface antigen (HBsAg) or hepatitis C (HCV) antibody
3. Known history of HIV infection
4. Known hypersensitivity to pilocarpine or pilocarpine-like muscarinic agonists
5. Known hypersensitivity to lidocaine or lidocaine-like agents
6. Presence of pacemakers
7. Subjects who are not able or are not willing to comply with the procedures of this protocol
8. Subject has a condition which in the opinion of the investigator would not allow for safe conduct of the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 42 days

SECONDARY OUTCOMES:
Exploratory endpoint: change from baseline in biological activity | Baseline and 42 days
  * Hair number and growth properties
  * Pulmonary function and eNO levels
  * Sweat duct density
  * Sweat rate
  * Saliva quantitation
  * Tearing and dry eye evaluation
  * Skin biopsy for expression profile

CONTACTS AND LOCATIONS:
Overall Officials: Ophir Klein, MD, PhD, Principal Investigator — University of California, San Francisco; James Maynard, MD, Principal Investigator — Community Research
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Community Research, Cincinnati, Ohio